CLINICAL TRIAL: NCT01134445
Title: Prospective, International Multi-centre, Uncontrolled, Post Marketing Surveillance Study to Monitor the Long-term Performance of the DePuy PROXIMA™ Hip in Subjects With Indications Suitable for a Primary Total Hip Arthroplasty
Brief Title: An Electronic Data Capture Study to Assess the Long-term Performance of the DePuy PROXIMA™ Hip in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated early for business reasons
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT07/02
Record Dates: First submitted 2010-03-05; First posted 2010-06-02 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Avascular Necrosis; Traumatic Femoral Fractures; Congenital Hip Dysplasia
Keywords: Arthroplasty; Replacement; Hip; Conservative; Anatomic; Cementless
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy Proxima™ Hip (Other): A short, anatomic, cementless femoral component for use in total hip arthroplasty
  Interventions: Device: DePuy Proxima™ Hip

INTERVENTIONS:
Device: DePuy Proxima™ Hip — A short, anatomic, cementless femoral component for use in total hip arthroplasty

SUMMARY:
The purpose of this study is to monitor the performance of the DePuy PROXIMA™ hip in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 70 years of age.
* Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and agree to return to the hospital for all the required post-operative follow-ups.
* Subjects who are scheduled to undergo a primary THR whom the surgeon considers to be suitable for the DePuy PROXIMATM hip femoral prosthesis.

Exclusion Criteria:

* Subjects with active local or systemic infection
* Subjects with loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
* Subjects with poor bone quality, such as osteoporosis, where, in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
* Subjects with Charcot's or Paget's disease.
* Subjects with hip dysplasia with severe neck anteversion or severe dysplasia of the proximal femur.
* Subjects with severe osteoporosis.
* Subjects with previous proximal femoral fractures.
* Subjects who, in the opinion of the Investigator, have an existing condition/co-morbidity or infection that would compromise their long-term participation and follow-up in this study.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).
* Subjects who are currently involved in any injury litigation claims.
* Subjects for whom the surgical procedure is a revision of a previous THR, hemi-arthroplasty or hip resurfacing
* Subjects who have previously undergone osteotomy or arthrodesis of the hip.
* Subjects undergoing a simultaneous bilateral hip operation.
* Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip is part of this clinical investigation.
* Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip was implanted less than six months previously or is not performing satisfactorily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the five-year time-point | 5yrs post surgery

SECONDARY OUTCOMES:
Annual Kaplan-Meier survivorship calculations | 1yr post-surgery
Harris Hip Score | 6mths post-surgery
Oxford Hip Score | 3mths post-surgery
UCLA Activity Score | 3mths post-surgery
Hip Outcome Score | 3mths post-surgery
EuroQol EQ-5D | 3mths post-surgery
Annual Kaplan-Meier survivorship calculations | 2yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 3yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 4yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 6yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 7yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 8yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 9yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 10yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 11yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 12yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 13yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 14yrs post-surgery
Annual Kaplan-Meier survivorship calculations | 15yrs post-surgery
Harris Hip Score | 1yr post-surgery
Harris Hip Score | 2yrs post-surgery
Harris Hip Score | 5yrs post-surgery
Harris Hip Score | 10yrs post-surgery
Harris Hip Score | 15yrs post-surgery
Radiographic Analysis | 3mths post-surgery
Radiographic Analysis | 6mths post-surgery
Radiographic Analysis | 1yr post-surgery
Radiographic Analysis | 2yrs post-surgery
Radiographic Analysis | 5yrs post-surgery
Radiographic Analysis | 10yrs post-surgery
Radiographic Analysis | 15 yrs post-surgery
Oxford Hip Score | 6mths post-surgery
Oxford Hip Score | 1yr post-sugery
UCLA Activity Score | 6mths post-surgery
UCLA Activity Score | 1yr post-surgery
Hip Outcome Score | 6mths post-surgery
Hip Outcome Score | 1yr post-surgery
EuroQol EQ-5D | 6mths post-surgery
EuroQol EQ-5D | 1yr post-surgery
Oxford Hip Score | 2yrs post-surgery
Oxford Hip Score | 3yrs post-surgery
Oxford Hip Score | 4yrs post-surgery
Oxford Hip Score | 5yrs post-surgery
Oxford Hip Score | 6yrs post-surgery
Oxford Hip Score | 7yrs post-surgery
Oxford Hip Score | 8yrs post-surgery
Oxford Hip Score | 9yrs post surgery
Oxford Hip Score | 10yrs post-surgery
Oxford Hip Score | 11yrs post-surgery
Oxford Hip Score | 12yrs post-surgery
Oxford Hip Score | 13yrs post-sugery
Oxford Hip Score | 14yrs post-surgery
Oxford Hip Score | 15yrs post-surgery
UCLA Activity Score | 2yrs post-surgery
UCLA Activity Score | 3yrs post-surgery
UCLA Activity Score | 4yrs post-surgery
UCLA Activity Score | 5yrs post-surgery
UCLA Activity Score | 6yrs post-surgery
UCLA Activity Score | 7yrs post-surgery
UCLA Activity Score | 8yrs post-surgery
UCLA Activity Score | 9yrs post-surgery
UCLA Activity Score | 10yrs post-surgery
UCLA Activity Score | 11yrs post-surgery
UCLA Activity Score | 12yrs post-surgery
UCLA Activity Score | 13yrs post-surgery
UCLA Activity Score | 14yrs post-surgery
UCLA Activity Score | 15yrs post-surgery
Hip Outcome Score | 2yrs post-surgery
Hip Outcome Score | 3yrs post-surgery
Hip Outcome Score | 4yrs post-surgery
Hip Outcome Score | 5yrs post-surgery
Hip Outcome Score | 6yrs post-surgery
Hip Outcome Score | 7yrs post-surgery
Hip Outcome Score | 8yrs post-surgery
Hip Outcome Score | 9yrs post-surgery
Hip Outcome Score | 10yrs post-surgery
Hip Outcome Score | 11yrs post-surgery
Hip Outcome Score | 12yrs post-surgery
Hip Outcome Score | 13yrs post-surgery
Hip Outcome Score | 14yrs post-surgery
Hip Outcome Score | 15yrs post-surgery
EuroQol EQ-5D | 2yrs post-surgery
EuroQol EQ-5D | 3yrs post-surgery
EuroQol EQ-5D | 4yrs post-surgery
EuroQol EQ-5D | 5yrs post-surgery
EuroQol EQ-5D | 6yrs post-surgery
EuroQol EQ-5D | 7yrs post-surgery
EuroQol EQ-5D | 8yrs post-surgery
EuroQol EQ-5D | 9yrs post-surgery
EuroQol EQ-5D | 10yrs post-surgery
EuroQol EQ-5D | 11yrs post-surgery
EuroQol EQ-5D | 12yrs post-surgery
EuroQol EQ-5D | 13yrs post-surgery
EuroQol EQ-5D | 14yrs post-surgery
EuroQol EQ-5D | 15yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Belle Isle, Metz, France
- Hospital de Santo Antonio, Porto, Portugal
- Hospital Clinic Barcelona, Barcelona, Spain
- Pilgrim Hospital, Boston, United Kingdom